CLINICAL TRIAL: NCT03126383
Title: Characterization of Inflammatory Muscle Involvement in Patients With Primary Sjögren's Syndrome
Brief Title: Inflammatory Myopathies in Primary Sjögren's Syndrome
Acronym: AMISS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: AMISS (29BRC17.0031)
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Primary Sjögren Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The AMISS study will characterize the features of muscle disease in patients with primary Sjogren's syndrome (pSS).

DETAILED DESCRIPTION:
Muscle disease is associated with pSS, but this association is not well defined. The AMISS study, a retrospective observational multicentric study, will recruit patients with pSS and muscle involvement in order to characterize in details the features of this association (epidemiological aspects, clinical presentation, biological, radiological and histological findings, treatments and outcomes).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Primary Sjögren's syndrome according to the ACR/EULAR classification criteria
* inflammatory muscle involvement, as diagnosed by the treating physician

Exclusion Criteria:

* Diagnosis of inflammatory myopathy before the diagnosis of pSS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Sjögren's syndrome
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-10 (Estimated); Primary Completion 2018-04-10 (Estimated); Study Completion 2018-04-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients fulfilling classification criteria for inflammatory myopathies | At diagnosis
  Among the patients included in the AMISS study, we will assess the proportion of patients who fulfill the classification criteria for the different inflammatory myopathies.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France